CLINICAL TRIAL: NCT06163859
Title: Female Community Health Volunteers Led Hypertension Prevention and Control in Nepal: An Implementation Study
Brief Title: Female Community Health Volunteers Led Hypertension Prevention and Control in Nepal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kathmandu University School of Medical Sciences (Other)
Collaborators: World Health Organization (Other); Institute for Implementation Science and Health (Unknown)
Responsible Party: Principal Investigator, Archana Shrestha, Professor, Kathmandu University School of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 459
Record Dates: First submitted 2023-11-16; First posted 2023-12-11 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Hypertension
Keywords: Community Health Workers; Hypertension Control; Hypertension Prevention; Implementation Study
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Female Community Health Volunteers (FHPC) implementation strategy
  Interventions: Behavioral: Intervention Group
- Control Arm (No Intervention): Routine hypertension care

INTERVENTIONS:
Behavioral: Intervention Group — FCHVs will undergo a 3-day training program on hypertension management, including screening, counseling, medication adherence, self-care, and referrals. FCHVs will form groups for individuals with hypertension and hold monthly meetings to discuss control strategies, review BP logs, and promote healthcare visits, including family involvement. They will also maintain regular communication with healthcare facility in-charges to ensure effective collaboration in the 'Hypertension Care Cascade Model'.
  Arms: Intervention Group

SUMMARY:
Brief Summary Hypertension is a major public health problem in Nepal, with substantial gaps in awareness, treatment, and control, particularly in rural and semi-urban settings. Nepal has adopted the WHO Package of Essential Non-Communicable Diseases (PEN) to strengthen facility-based hypertension care; however, persistent community- and system-level barriers limit its effectiveness.

This study evaluates a Female Community Health Volunteer (FCHV)-led, community-based hypertension prevention and control intervention in Namobuddha Municipality, Kavrepalanchowk District, Nepal. The study uses a hybrid type II effectiveness-implementation cluster randomized controlled trial design to assess both implementation outcomes and clinical effectiveness. Twelve public primary healthcare facilities are randomized (1:1) to intervention or routine care. Implementation outcomes are assessed using the RE-AIM framework (Reach, Effectiveness, Adoption, and Implementation). The primary effectiveness outcome is change in mean systolic blood pressure at three months. Secondary outcomes include diastolic blood pressure, hypertension control status, hypertension knowledge, dietary behavior, medication adherence, and body mass index. The intervention mobilizes trained FCHVs to deliver group-based blood pressure monitoring, structured health education, lifestyle counseling, medication adherence support, and referral linkages to primary healthcare facilities.

DETAILED DESCRIPTION:
Study design: The investigators will conduct a Hybrid type II effectiveness-implementation design focusing on implementation outcomes while also collecting effectiveness outcomes as they relate to the uptake or fidelity of the intervention. A mixed-method approach will be used. The investigators will conduct a cluster randomized controlled trial among 520 participants, clustered within 12 health facilities. Among the participants of the intervention arm, the investigators will collect quantitative data on adoption, implementation and reach. The investigators will conduct in-depth interviews with 8-16 patients, at least 2 FGDs with FCHVs and at least 4 Key Informant Interviews (KIIs) with health workers to understand implementation outcomes. The investigators will maintain qualitative tracking logs to document meetings with FCHVs and healthcare workers.

Study site: In partnership with the Ministry of Health and Population (MoHP), the World Health Organization (WHO), and the NCD Flagship Initiative, and with funding from the Norwegian government, Bagmati province has initiated the Hypertension care cascade model in the Kavrepalnchowk district. In this context, our research aims to support the model's objectives by monitoring treatment outcomes and control rates at every stage of care in the Kavre district. The study will involve 12 basic health facilities in Namobuddha municipalities of Kavrepalnchowk, where approximately 82 female community health volunteers (FCHVs) are actively engaged. The selection of the study district and municipalities was done in consultation with WHO Nepal and Nepal Health Research Council, taking into consideration national priorities, Norad priorities, and ongoing NCD care activities in the district.

Study Population: At the facility level, the investigators will include basic health facilities that have implemented PEN, excluding those who are not within the network of the Nepal government health system. At the patient level, inclusion criteria will be: i) 30-75 years old ii) have a high blood pressure of 130/80 mmHg, iii) are able to provide informed consent. Exclusion criteria will include: severe illness requiring bed-rest, and pregnant women due to their special health needs.

Intervention :

We propose a community-based hypertension intervention in Namobuddha Municipality, leveraging Female Community Health Volunteers (FCHVs) as frontline implementers. A total of 34 FCHVs will each form a group of 7-16 participants and conduct one-hour, bi-monthly sessions over three months. Sessions will include:

Blood pressure monitoring Structured health education on hypertension and its risk factors Counseling on lifestyle modification Support for medication adherence Referral to primary care for participants with uncontrolled blood pressure

FCHVs are selected due to their trusted status and strong community presence, which facilitate participant engagement and behavior change. Evidence from Nepal and other settings demonstrates that community health workers are effective agents for hypertension prevention and control. Regular blood pressure monitoring raises awareness and promotes timely care-seeking, while structured education grounded in Social Cognitive Theory enhances knowledge, self-efficacy, and peer-supported behavior change . The group-based delivery model integrates behavioral and clinical interventions in a low-cost, sustainable framework.

Implementation Strategies

Implementation will follow an Implementation Research Logic Model (IRLM) to align strategies, mechanisms, and expected outcomes. Development of these strategies included:

Consultations with health workers and municipal health coordinators Cognitive interviews with FCHVs from neighboring municipalities Meetings with federal, provincial, and local government authorities These consultations informed locally adapted intervention materials, including flip charts and other literacy-appropriate tools, designed to match FCHVs' skills, workload, and the sociocultural context.

The implementation strategies are designed to address key barriers and leverage facilitators identified during formative assessments and prior evidence on FCHV-led interventions:

Capacity Building: A one-time, three-day competency-based training to strengthen FCHVs' skills in blood pressure measurement, behavior change communication, documentation, and goal setting.

Technical and Clinical Support: Provision of digital automated blood pressure monitors and literacy-appropriate materials to enable accurate measurement and effective education delivery.

Coalition Building: Formation of FCHV-led hypertension groups meeting twice monthly to support lifestyle changes, medication adherence, and self-care.

Community-Facility Linkages: Monthly coordination and referral meetings between FCHVs and health facility in-charges to strengthen referral systems, enhance communication, and create feedback loops for problem-solving.

Tools and data collection: Quantitative data will be collected using face-to-face interviews administered by trained research assistants using standardized questionnaires adapted from the WHO STEPS survey , Hypertension Knowledge, Hill bone compliance , Dietary quality questionnaire and entered into REDCap. Blood pressure will be measured using a standardized protocol. Qualitative data will be collected through supportive process documentation to inform interpretation of implementation outcomes.

Blood pressure will be taken during baseline and endline. The investigators will be using both quantitative and qualitative tools to measure our primary outcomes. The investigators will conduct In-depth interviews (IDIs) and Focus group discussion (FGDs) and transcribe all the discussions and interviews into Nepali. The principal investigators and local principal investigator then independently review the transcripts against the audio recording for potential discrepancies or incomplete data. The investigators will conduct abductive analysis, using first inductive codes (e.g., emerging from the data) and transposing these into deductive REAIM domain. RAs will keep field notebooks to document observed behaviors of providers and patients relevant to implementation.

For qualitative information collection, the investigators will develop an IDI guide based on previous literature for qualitative study.

Data analysis:

1. The investigators will compute estimates of adoption, implementation, reach and maintenance, with appropriate 95% confidence intervals. Reach is defined as % of FCHVs implementing the program will participate in monthly meetings; at Client level: percent of the hypertensive patients in the community are aware of their high BP status. Adoption is defined as % of the health facilities asked to participate in adopting the program i.e. FCHVs complete the initial training session. Program implementation is defined as % of the health facility will implement a minimum standard to program implementation, measured by: (1) healthcare workers conduct monthly meetings; (2) first home visits by FCHVs to the target clients; and (3) FCHV submit monthly reports. In addition, the investigators will explore facilitators and barriers to implementation.
2. For qualitative FGDs and interviews, the investigators will conduct abductive analysis36, using first inductive codes (e.g., emerging from the data) and transposing these into deductive CFIR constructs. RAs will keep field notebooks to document observed behaviors of providers and patients relevant to implementation.
3. The baseline characteristics will be presented as the mean (standard deviation) or, median (interquartile) for continuous; and frequency (%) for categorical variables. Primary analyses of the outcome, mean systolic BP at 3 months using paired t-test.

The investigators will conduct a mixed-methods assessment of the implementation outcomes by combining data from quantitative tools and from in-depth interviews.

ELIGIBILITY:
Inclusion Criteria:

* 30 -75 years old
* have a high blood pressure of 130/80 mmHg or under hypertension medication
* are able to provide informed consent.

Exclusion Criteria:

* severe illness requiring bed rest, and
* pregnant women, due to their special health needs.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2025-03-16 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Reach | 3 months
  The proportion of the target population that participates in the intervention.
  Indicators: Proportion of individuals screened during one-day hypertension screening camps in each health facilities by FCHVs.( denomiator will be determined using national prevalence of hypertension).
  Data Source: Patient records maintained by FCHV, attendance sheets from FCHV-HTN group meetings.
  Demographic distribution (age, gender, etc.) of the individuals screened.
Adoption | 3 months
  Adoption is defined as the proportion of eligible health facilities that agreed to participate in the study. Participation will be confirmed through signed minutes from meetings between the municipal health coordinator and facility representatives, indicating formal approval to implement the program.
Implementation | 3 months
  The extent to which the FCHV-led intervention is delivered as intended.
  Indicators: Number of FCHVs conducting complete (3 months) FCHV-HTN meetings, Documentation and follow-up of participants' blood pressure logs by FCHVs, duration of sessions conducted, number of sessions conducted.
  Data source: Forms sent by FCHV at health facilities (compiled at Health facilities), logs maintained by FCHVs
Mean systolic blood pressure (BP) (mmHg) | 3 months
  The net change in mean systolic BP between intervention and control

SECONDARY OUTCOMES:
Mean diastolic BP (mmHg) | 3 months
  Net change in mean diastolic BP from baseline to follow up
Physical activity | 3 months
  The proportion engaged in moderate physical activity (2.5 hours per week) measured at baseline and follow up
Fruits and vegetables intake | 3 months
  The proportion consuming diet high in fruits and vegetables in the last 24 hours self reported at baseline and follow up
Medication adherence | 3 months
  The proportion adhering to prescribed medication in the past two weeks measured at baseline and follow up
Proportion controlling BP (<140/90 mmHg) | 3 months
  Proportion of participants controlling BP (<140/90 mmHg) from baseline to follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Implementation Science and Health, Kavre, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopez AD, Mathers CD, Ezzati M, Jamison DT, Murray CJ. Global and regional burden of disease and risk factors, 2001: systematic analysis of population health data. Lancet. 2006 May 27;367(9524):1747-57. doi: 10.1016/S0140-6736(06)68770-9. PMID 16731270
- [Background] Aryal KK, Mehata S, Neupane S, Vaidya A, Dhimal M, Dhakal P, Rana S, Bhusal CL, Lohani GR, Paulin FH, Garg RM, Guthold R, Cowan M, Riley LM, Karki KB. The Burden and Determinants of Non Communicable Diseases Risk Factors in Nepal: Findings from a Nationwide STEPS Survey. PLoS One. 2015 Aug 5;10(8):e0134834. doi: 10.1371/journal.pone.0134834. eCollection 2015. PMID 26244512
- [Background] Karmacharya BM, Koju RP, LoGerfo JP, Chan KC, Mokdad AH, Shrestha A, Sotoodehnia N, Fitzpatrick AL. Awareness, treatment and control of hypertension in Nepal: findings from the Dhulikhel Heart Study. Heart Asia. 2017 Jan 4;9(1):1-8. doi: 10.1136/heartasia-2016-010766. eCollection 2017. PMID 28123454
- [Background] Sacks FM, Svetkey LP, Vollmer WM, Appel LJ, Bray GA, Harsha D, Obarzanek E, Conlin PR, Miller ER 3rd, Simons-Morton DG, Karanja N, Lin PH; DASH-Sodium Collaborative Research Group. Effects on blood pressure of reduced dietary sodium and the Dietary Approaches to Stop Hypertension (DASH) diet. DASH-Sodium Collaborative Research Group. N Engl J Med. 2001 Jan 4;344(1):3-10. doi: 10.1056/NEJM200101043440101. PMID 11136953
- [Background] Svetkey LP, Simons-Morton DG, Proschan MA, Sacks FM, Conlin PR, Harsha D, Moore TJ. Effect of the dietary approaches to stop hypertension diet and reduced sodium intake on blood pressure control. J Clin Hypertens (Greenwich). 2004 Jul;6(7):373-81. doi: 10.1111/j.1524-6175.2004.03523.x. PMID 15249792
- [Background] Parker ED, Schmitz KH, Jacobs DR Jr, Dengel DR, Schreiner PJ. Physical activity in young adults and incident hypertension over 15 years of follow-up: the CARDIA study. Am J Public Health. 2007 Apr;97(4):703-9. doi: 10.2105/AJPH.2004.055889. Epub 2007 Feb 28. PMID 17329668
- [Background] Ascherio A, Hennekens C, Willett WC, Sacks F, Rosner B, Manson J, Witteman J, Stampfer MJ. Prospective study of nutritional factors, blood pressure, and hypertension among US women. Hypertension. 1996 May;27(5):1065-72. doi: 10.1161/01.hyp.27.5.1065. PMID 8621198
- [Background] Zachariah R, Ford N, Philips M, Lynch S, Massaquoi M, Janssens V, Harries AD. Task shifting in HIV/AIDS: opportunities, challenges and proposed actions for sub-Saharan Africa. Trans R Soc Trop Med Hyg. 2009 Jun;103(6):549-58. doi: 10.1016/j.trstmh.2008.09.019. Epub 2008 Nov 6. PMID 18992905
- [Background] Jindal D, Sharma H, Gupta Y, Ajay VS, Roy A, Sharma R, Ali M, Jarhyan P, Gupta P, Srinivasapura Venkateshmurthy N, Ali MK, Narayan KMV, Prabhakaran D, Weber MB, Mohan S, Patel SA, Tandon N. Improving care for hypertension and diabetes in india by addition of clinical decision support system and task shifting in the national NCD program: I-TREC model of care. BMC Health Serv Res. 2022 May 23;22(1):688. doi: 10.1186/s12913-022-08025-y. PMID 35606762
- [Background] Labhardt ND, Balo JR, Ndam M, Grimm JJ, Manga E. Task shifting to non-physician clinicians for integrated management of hypertension and diabetes in rural Cameroon: a programme assessment at two years. BMC Health Serv Res. 2010 Dec 14;10:339. doi: 10.1186/1472-6963-10-339. PMID 21144064
- [Background] Sun Y, Mu J, Wang DW, Ouyang N, Xing L, Guo X, Zhao C, Ren G, Ye N, Zhou Y, Wang J, Li Z, Sun G, Yang R, Chen CS, He J; CRHCP Study Group. A village doctor-led multifaceted intervention for blood pressure control in rural China: an open, cluster randomised trial. Lancet. 2022 May 21;399(10339):1964-1975. doi: 10.1016/S0140-6736(22)00325-7. Epub 2022 Apr 29. PMID 35500594
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Neupane D, McLachlan CS, Mishra SR, Olsen MH, Perry HB, Karki A, Kallestrup P. Female community health volunteers to reduce blood pressure: feasible and sustainable? - Authors' reply. Lancet Glob Health. 2018 Apr;6(4):e374. doi: 10.1016/S2214-109X(18)30033-0. No abstract available. PMID 29530417
- [Background] Neupane D, McLachlan CS, Mishra SR, Olsen MH, Perry HB, Karki A, Kallestrup P. Effectiveness of a lifestyle intervention led by female community health volunteers versus usual care in blood pressure reduction (COBIN): an open-label, cluster-randomised trial. Lancet Glob Health. 2018 Jan;6(1):e66-e73. doi: 10.1016/S2214-109X(17)30411-4. PMID 29241617
- [Background] Gearing RE, El-Bassel N, Ghesquiere A, Baldwin S, Gillies J, Ngeow E. Major ingredients of fidelity: a review and scientific guide to improving quality of intervention research implementation. Clin Psychol Rev. 2011 Feb;31(1):79-88. doi: 10.1016/j.cpr.2010.09.007. Epub 2010 Oct 7. PMID 21130938
- [Background] Shrestha A, Maharjan R, Karmacharya BM, Bajracharya S, Jha N, Shrestha S, Aryal A, Baral PP, Bhatt RD, Bhattarai S, Bista D, Citrin D, Dhimal M, Fitzpatrick AL, Jha AK, Karmacharya RM, Mali S, Neupane T, Oli N, Pandit R, Parajuli SB, Pradhan PMS, Prajapati D, Pyakurel M, Pyakurel P, Rai BK, Sapkota BP, Sapkota S, Shrestha A, Shrestha AP, Shrestha R, Sharma GN, Sharma S, Spiegelman D, Suwal PS, Thapa B, Vaidya A, Xu D, Yan LL, Koju R. Health system gaps in cardiovascular disease prevention and management in Nepal. BMC Health Serv Res. 2021 Jul 5;21(1):655. doi: 10.1186/s12913-021-06681-0. PMID 34225714
- See also: World Health Organization, Ministry of Health and Population. Multisectoral Action Plan for the Prevention and Control of Non Communicable Diseases (2014-2020) — http://who.int/docs/default-source/nepal-documents/multisectoral-action-plan-for-prevention-and-control-of-ncds-(2014-2020).pdf?sfvrsn=c3fa147c_4